CLINICAL TRIAL: NCT02160470
Title: Enhancing Exposure Therapy for Snake and Spider Phobias With Fear Retrieval and Compound Extinction
Brief Title: Enhancing Exposure Therapy for Snake and Spider Phobias
Acronym: Snake/Spider
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Texas at Austin (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Michael J. Telch, Professor, University of Texas at Austin
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: 2011-10-0012; 1F31MH100760-01 (NIH)
Record Dates: First submitted 2014-01-22; First posted 2014-06-10 (Estimated); Last update posted 2020-12-08 (Actual); Status verified 2020-12

CONDITIONS: Specific Phobia
MeSH Terms: conditions — Phobia, Specific | interventions — Implosive Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Exposure with Retrieval (Experimental): Exposure Therapy with Retrieval
  Interventions: Behavioral: Exposure Therapy with Retrieval
- Exposure with Compounding (Experimental): Exposure Therapy with Compound Extinction
  Interventions: Behavioral: Exposure Therapy with Compound Extinction
- Exposure with Retrieval and Compounding (Experimental): Exposure Therapy with Retrieval and Compound Extinction
  Interventions: Behavioral: Exposure Therapy with Retrieval and Compound Extinction
- Therapist-Guided Exposure Therapy (Active Comparator): Therapist-guided Exposure Therapy
  Interventions: Behavioral: Therapist-guided Exposure Therapy

INTERVENTIONS:
Behavioral: Exposure Therapy with Retrieval — Participants will receive one-session exposure therapy (up to 92 minutes) for fear of spiders or fear of snakes. Thirty minutes prior to exposure therapy, participants will receive a fear retrieval trial, which is a brief exposure to the feared stimulus (snake or spider). Based on recent basic science research, the fear retrieval trial is expected to enhance the efficacy of exposure therapy.
  Arms: Exposure with Retrieval
Behavioral: Exposure Therapy with Compound Extinction — Participants will receive one-session exposure therapy (up to 92 minutes) for fear of spiders or fear of snakes. As a component of therapy, participants will receive compound extinction, which consists of exposure to two feared stimuli simultaneously (two spiders or two snakes). Based on recent basic science research, compound extinction is expected to enhance the efficacy of exposure therapy.
  Arms: Exposure with Compounding
Behavioral: Exposure Therapy with Retrieval and Compound Extinction — Participants will receive one-session exposure therapy (up to 92 minutes) for fear of spiders or fear of snakes. Thirty minutes prior to exposure therapy, participants will receive a brief fear retrieval trial. As a component of therapy, participants will also receive compound extinction.
  Arms: Exposure with Retrieval and Compounding
Behavioral: Therapist-guided Exposure Therapy — Participants will receive one-session exposure therapy (up to 92 minutes) for fear of spiders or fear of snakes.
  Arms: Therapist-Guided Exposure Therapy

SUMMARY:
This study tests whether exposure therapy for fear of snakes or spiders is enhanced by the addition of a brief fear retrieval trial prior to treatment, and the use of compound extinction during treatment. The goal of the study is to determine whether these behavioral techniques enhance the efficacy of exposure therapy, one of the most empirically supported treatments for anxiety disorders.

DETAILED DESCRIPTION:
This study tests whether exposure therapy for fear of snakes or spiders is enhanced by the addition of a brief fear retrieval trial prior to treatment, and the use of compound extinction during treatment. The goal of the study is to determine whether these behavioral techniques enhance the efficacy of exposure therapy, one of the most empirically supported treatments for anxiety disorders. Individuals between the ages of 18-65 with elevated fear of spiders or fear of snakes are randomly assigned to one of four treatment conditions (1) standard exposure therapy, (2) exposure therapy with fear retrieval augmentation, (3) exposure therapy with compound extinction augmentation, and (4) exposure therapy with fear retrieval and compound extinction augmentations. All participants undergo an online prescreen and a face-to-face screening assessment to determine eligibility and baseline (pre-treatment) symptom severity. Participants additionally complete assessments directly after treatment (post-treatment), and approximately one week after treatment (follow-up). The pre-treatment assessment occurs 1-14 days prior to treatment, the post-treatment assessment occurs during the treatment visit as soon as the treatment procedure is complete, and the follow-up assessment occurs within a window of 6-14 days after the completion of treatment. Participants complete two behavioral approach tests (in the treatment context and in the generalization context) at pre-treatment, post-treatment, and follow-up. Participants complete a battery of self-report questionnaires at pre-treatment and follow-up.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 to 65.
2. Speaks English fluently.
3. A score of 70 or higher on the Fear of Snakes/Spiders Questionnaire.
4. Demonstrates avoidance during behavioral approach tests (defined as inability to put palm flat on the bottom of a tank containing a snake/spider, and inability to touch a snake/spider with a bare finger).

Exclusion Criteria:

1. Unstable dose of psychotropic medications during the 4 weeks prior to baseline assessment.
2. Currently receiving exposure-based treatment for snake/spider phobia.
3. Currently at risk for suicide.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2012-08 (Actual); Primary Completion 2019-12 (Actual); Study Completion 2019-12 (Actual)

PRIMARY OUTCOMES:
Change in peak subjective fear (0 - 100), behavioral approach (0 - 4), and heart rate reactivity to a live snake/spider not used during treatment (generalization context) from pre-treatment to follow-up | pre-treatment (window of 1-14 days prior to treatment); follow-up (window of 6-14 days after treatment)

SECONDARY OUTCOMES:
Change in peak subjective fear (0 - 100), behavioral approach (0 - 4), and heart rate reactivity to a live snake/spider not used during treatment (generalization context) from pre-treatment to post-treatment. | pre-treatment (window of 1-14 days prior to treatment); post-treatment (directly after the treatment procedure is completed)
Change in peak subjective fear (0 - 100), behavioral approach (1 - 8), and heart rate reactivity to a live snake/spider used during treatment (treatment context) from pre-treatment to follow-up | pre-treatment (window of 1-14 days prior to treatment); follow-up (window of 6-14 days after treatment)
Change in peak subjective fear (0 - 100), behavioral approach (1 - 8), and heart rate reactivity to a live snake/spider used during treatment (treatment context) from pre-treatment to post-treatment | pre-treatment (window of 1-14 days prior to treatment); post-treatment (directly after the treatment procedure is completed)
Change in Fear of Snakes/Spiders Questionnaire from pre-treatment to follow-up | pre-treatment (window of 1-14 days prior to treatment); follow-up (window of 6-14 days after treatment)
Change in Snake/Spider Belief Questionnaire from pre-treatment to follow-up | pre-treatment (window of 1-14 days prior to treatment); follow-up (window of 6-14 days after treatment)
Change in Agoraphobic Cognitions Questionnaire for Snake/Spider Phobia from pre-treatment to follow-up | pre-treatment (window of 1-14 days prior to treatment); follow-up (window of 6-14 days after treatment)
Change in Self-Efficacy Questionnaire for Spider/Snake Phobia from pre-treatment to follow-up | pre-treatment (window of 1-14 days prior to treatment); follow-up (window of 6-14 days after treatment)
Change in Armfield and Mattiske Disgust Questionnaire from pre-treatment to follow-up | pre-treatment (window of 1-14 days prior to treatment); follow-up (window of 6-14 days after treatment)
Change in Lab for the Study of Anxiety Disorders Specific Phobia Diagnostic Questionnaire from pre-treatment to follow-up | pre-treatment (window of 1-14 days prior to treatment); follow-up (window of 6-14 days after treatment)
  change from pre-treatment in current phobic diagnostic status and in level of phobic-related distress and impairment

CONTACTS AND LOCATIONS:
Overall Officials: Michael J Telch, PhD, Principal Investigator — University of Texas at Austin
Locations (1):
- University of Texas at Austin, Austin, Texas, United States

REFERENCES:
- [Derived] Lancaster CL, Monfils MH, Telch MJ. Augmenting exposure therapy with pre-extinction fear memory reactivation and deepened extinction: A randomized controlled trial. Behav Res Ther. 2020 Dec;135:103730. doi: 10.1016/j.brat.2020.103730. Epub 2020 Sep 19. PMID 33096291